CLINICAL TRIAL: NCT01801592
Title: Prevalence of Obstructive Sleep Apnoea in Patients With Intermittent Claudication
Brief Title: Obstructive Sleep Apnoea in Patients With Intermittent Claudication
Acronym: WITH-SAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2012-A01124-39
Record Dates: First submitted 2013-02-18; First posted 2013-03-01 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2016-02

CONDITIONS: Sleep Apnea
Keywords: OBSTRUCTIVE SLEEP APNOEA; INTERMITTENT CLAUDICATION; Respiratory disease; Peripheral artery disease
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Intermittent Claudication; Respiration Disorders; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main aim of this study is to determine how common undiagnosed obstructive sleep apnoea is in individuals with intermittent claudication.

DETAILED DESCRIPTION:
In patients with peripheral artery disease (PAD), exercise induced limb ischemia (claudication) which limits walking capacity. Symptoms are due to pain at hip and/or buttock. Couple of origins may induce this pain such as vascular, cardiac, respiratory, musculoskeletal, neurologic, hematologic etc. The rate of associated respiratory pathology to patients with lower extremity artery disease (LEAD) is around 15%. The intolerance to walk could be link to an exercise hypoxia which appears with lower limb pain with or without associated dyspnea. The exercise hypoxemia becomes a diagnostic for an intermittent vascular claudication. Tests which are performed to diagnose an intermittent claudication are the Ankle to Brachial Systolic pressure Index (ABI), the echo-Doppler of lower limb arteries and the walking test on a treadmill associated to a measurement of the distal and chest transcutaneous oxygen pressure (tcpO2).

Thus, the purpose of the present research is to determine the prevalence of obstructive sleep apnoea in patient with PAD.

ELIGIBILITY:
Inclusion Criteria:

* Register to the social health insurance
* Referred for a walk test because of claudication
* Maximal walking ditance < 750m
* Older than 18 years old
* Able to understand the protocol of the study

Exclusion Criteria:

* Cardiac insufficiency already known, stage III or IV i.e. dyspnea at rest Unstable angina or myocardial infarction within the previous three months inclusion
* Severe reparatory disease already known
* Parkinson disease, hémiplégia ou paraplégia
* Does not want to participate to the protocol
* Pregnant women
* Adults to enhanced protection, deprived of their liberty by judicial or administrative authority, without consent hospitalized or admitted to a health facility or social purposes other than research
* Being in a period of exclusion from another biomedical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men or women over 18 years old with an Intermitent claudication.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2013-05-03 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Prevalence of an Apnea hyponea index > 15 | up to 2 months after inclusion
  Recording of sleep with the RESMED (Apnealink) system

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Mahe, MD; PhD, Principal Investigator — University Hospital in Angers
Locations (1):
- University hospital, Angers, France